CLINICAL TRIAL: NCT02406729
Title: Phase III, Double-Blind, Randomized, Placebo-Controlled Trial to Evaluate the Efficacy, Safety, and Immunogenicity of the Dengue 1, 2, 3, 4 (Attenuated) Vaccine From Instituto Butantan
Brief Title: Phase III Trial to Evaluate Efficacy and Safety of a Tetravalent Dengue Vaccine
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEN-03-IB; U1111-1168-8679 (Registry Identifier: UTN)
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dengue 1,2,3,4 (attenuated) vaccine (Experimental): Dengue 1,2,3,4 (attenuated) vaccine Single dose, SC
  Interventions: Biological: Dengue 1,2,3,4 (attenuated) vaccine
- Placebo (Placebo Comparator): Placebo Single dose, SC
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Dengue 1,2,3,4 (attenuated) vaccine — Dose 1000 PFU per virus (1,2,3,4) Route:subcutaneous
  Other Names: Butantan DV; TetraVax-DV-TV003
  Arms: Dengue 1,2,3,4 (attenuated) vaccine
Other: Placebo — Route:subcutaneous
  Arms: Placebo

SUMMARY:
This is a randomized, multicenter, double-blind, placebo-controlled Phase III study that will evaluate efficacy and safety of a live attenuated, tetravalent, lyophilized dengue vaccine produced by Butantan Institute.

The study will be carried out in multiple sites in Brazil. The study will be community-based in select urban areas where there's dengue transmission.

Study's intervention will be a single dose of the tetravalent dengue vaccine or placebo in a ratio 2:1. For efficacy analysis will be considered all dengue cases occurring after 28 days post-vaccination in the entire population of 16944 participants.

For safety analysis participants will be divided in three age groups: 18 to 59 ys, 7-17 ys and 2 to 6 ys. In each of these age groups there will be a minimum of 4992 participants. The age groups of 18 to 59 ys and 7 to 17 ys will start first. Once safety data for the first 21 days after vaccination is analysed for 450 participants in 7-to17-ys age group, the following group, of 2 to 6 ys, will start.

The study's hypothesis is that the vaccine under investigation and produced by Butantan Institute is safe and provides protection against dengue symptomatic disease of 80% or more with a lower bound of the 95% confidence interval of 25%. This way, the expected number of dengue cases virologically confirmed is 24 or more which will provide a response in terms of vaccine efficacy.

All participants will be followed up for five years to verify dengue incidence, regardless severity.

ELIGIBILITY:
Inclusion Criteria:

1. Children who have completed 24 months of age, adolescents and adults who have not completed 60 years of age;
2. Agree with periodic contacts, either/or by phone, electronic means, and home visits.
3. Show voluntary intention to participate in the study, documented by the participant's or participant's legal representative's signature of the informed consent form.

Exclusion Criteria:

1. For women: Pregnancy (confirmed by positive beta-hCG test) or breastfeeding;
2. Evidence of active neurological, cardiac, pulmonary, hepatic or renal disease as per clinical history and/or physical examination;
3. Compromised immune system diseases including: decompensated diabetes mellitus, cancer (except basal cell carcinoma), congenital or acquired immune deficiencies and not controlled autoimmune, as per clinical history and/or physical examination;
4. Behavioral, cognitive or psychiatric disease that in the opinion of the principal investigator or his representative physician, affects the participant ability to understand and cooperate with all study protocol requirements;
5. Abusive usage of alcohol or drugs in the past 12 months that has caused medical, professional or family problems, indicated by clinical history;
6. History of severe allergic reactions or anaphylaxis to the vaccine or to components of the vaccine in study;
7. History of asplenia;
8. Use of any investigational product within 28 days before or after receiving this study vaccination;
9. Has participated in another clinical trial six months prior to inclusion in the study or planning to participate in another clinical trial within 2 years following inclusion;
10. Use of immunosuppressant drugs such as: antineoplastic chemotherapy, radiation therapy, immunosuppressants to induce tolerance to transplants, and corticosteroids use (except topical or nasal). For this protocol will be considered for exclusion use of corticosteroids 3 months prior to the inclusion in the study and 6 months prior to the inclusion for the other therapies mentioned, and planned use of any immunosuppressant therapy within 2 years following inclusion in the study. It will be considered immunosuppressive dose of corticosteroids the equivalent to a dose ≥20 mg of prednisone per day for adults and the equivalent of prednisone at 2 mg/kg/day for children for over 7 days;
11. Have received blood products in the past three months, including transfusions or immunoglobulin, or scheduled administration of blood products or immunoglobulin for the following 2 years after vaccination;
12. Fever or suspected fever within 72 hours prior to vaccination or axillary temperature greater than 37,8°C on the day of vaccination (inclusion might be postponed until participant has completed 72 hours of no fever);
13. Have received live virus vaccine within 28 days or killed virus vaccine in the last 14 days prior to vaccination, or have a scheduled immunization during the first 28 days after receiving the investigational product;
14. Any other condition that might put in risk the safety/rights of a potential participant or hurdle his/her compliance with this protocol in investigator's opinion or his representative physician.

Ages: 24 Months to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16935 (Estimated)
Dates: Start 2016-02-22 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy (incidence density of symptomatic dengue cases, virologically confirmed) | Five years post vaccination, all cases after 28 days post-vaccination
  The primary efficacy outcome is incidence density of symptomatic dengue cases, virologically confirmed, after 28 days post-vaccination. Virological confirmation might be done by viral isolation, RT-PCR and/or detection of NS1.
Safety (adverse reactions) | In the first 21 days post-vaccination
  The primary safety outcome is the frequency of local and systemic adverse reactions, solicited and non-solicited in the three age groups, within the first 21 days post-vaccination. Adverse reactions are defined as adverse events that have a reasonable causal relationship with vaccination.

SECONDARY OUTCOMES:
Efficacy (incidence density of dengue cases confirmed virologically, regarding previous exposure to dengue viruses. ) | at five years post vaccination, all cases after 28 days post-vaccination
  The incidence density of dengue cases confirmed virologically after 28 days of vaccination, regarding previous exposure to dengue viruses. To demonstrate previous exposure or not to dengue viruses, validated serological methods such as: Elisa IgG Indirect, hemagglutination inhibition test or neutralizing antibodies (e.g., VRNT) or another validated test will be used. In case of doubtful results, more than one technique may be used to confirm the diagnosis.
Efficacy (incidence density of dengue cases confirmed virologically, regarding the viral serotype) | Five years post vaccination, all cases after 28 days post-vaccination
  The incidence density of dengue cases confirmed virologically after 28 days of vaccination, regarding the viral serotype. Virological diagnosis of the viral serotype will be performed using the viral isolation technique or RT-PCR.
Efficacy (incidence density of cases of severe dengue and/or with alarm signs, including cases hospitalized or not) | Five years post vaccination, all cases after 28 days post-vaccination
  Incidence density of cases of severe dengue and/or with alarm signs, including cases hospitalized or not, after 28 days of vaccination. Laboratory confirmation of these cases will occur through serological and/or virological tests.
Safety ( frequency of solicited and unsolicited local and systemic adverse reactions in participants regarding previous exposure to dengue viruses ) | In the first 21 days post-vaccination
  The frequency of solicited and unsolicited local and systemic adverse reactions in participants regarding previous exposure to dengue viruses during the 21-day period after vaccination.
Safety (frequency of unsolicited adverse reactions) | Five years post vaccination, all cases after the first 21 days post-vaccination
  The frequency of unsolicited adverse reactions after 21 days of vaccination until the end of the study.
Immunogenicity (consistency of the immune response to different batches of the vaccine ) | 4 weeks post vaccination
  The geometric mean of neutralizing antibody titers for each serotype in the fourth week after vaccination in a subgroup of adult participants without previous exposure to dengue immunized with three consecutive batches of dengue vaccine 1,2,3,4 (attenuated).
Immunogenicity (non-inferiority between simplified formulation vs. conventional formulation) | 4 weeks post vaccination
  The geometric mean of titers of neutralizing antibodies for each serotype at Week 4 postvaccination in a subgroup of adult participants without previous prior exposure to dengue and vaccinated with the conventional formulation and the simplified formulation of the dengue 1, 2, 3, 4 (attenuated) vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda C Boulos, MD, PhD, Study Director — Instituto Butantan
Locations (17):
- Brazil (17):
  - Fundação de Medicina Tropical Doutor Heitor Vieira Dourado, Manaus, Amazonas
  - Universidade Federal do Ceará, Fortaleza, Ceará
  - Instituto Gonçalo Muniz - Fiocruz Bahia, Simões Filho, Estado de Bahia
  - Universidade de Brasília, Brasília, Federal District
  - Universidade Federal de Mato Grosso do Sul, Campo Grande, Mato Grosso do Sul
  - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital Universitário Júlio Müller da Universidade Federal de Mato Grosso, Cuiabá, Mount
  - Centro de Pesquisas Aggeu Magalhães - Fiocruz Pernambuco, Recife, Pernambuco
  - Hospital Escola da Universidade Federal de Pelotas (HEUFPel), Pelotas, Rio Grande do Sul
  - Hospital São Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas em Medicina Tropical de Rondônia (CEPEM), Porto Velho, Rondônia
  - Universidade Federal de Roraima - UFRR, Boa Vista, Roraima
  - Universidade Federal de Sergipe, Laranjeiras, Sergipe
  - Faculdade de Medicina de São José do Rio Preto - FAMERP, São José do Rio Preto, São Paulo
  - Santa Casa de Misericórdia de São Paulo - CSEBF, São Paulo, São Paulo
  - Instituto de Infectologia Evandro Chagas - Fiocruz, Rio de Janeiro
  - HCFMUSP, São Paulo

REFERENCES:
- [Background] Precioso AR, Palacios R, Thome B, Mondini G, Braga P, Kalil J. Clinical evaluation strategies for a live attenuated tetravalent dengue vaccine. Vaccine. 2015 Dec 10;33(50):7121-5. doi: 10.1016/j.vaccine.2015.09.105. Epub 2015 Oct 14. PMID 26458796
- [Derived] Peixoto de Miranda EJF, de Sousa Moreira JA, da Silva Braga R, Silveira DHR, Infante V, de Oliveira Alves LB, de Camargo Vieira Tenorio J, Dos Santos Silva GF, Patino EG, de Mesquita Pacheco PHT, Ramos F, Oliveira DS, Kallas EG, Boulos FC. Randomized, double-blind, placebo-controlled, phase 3 trial to demonstrate lot-to-lot consistency of 3 lots of the simplified formulation of Butantan-dengue vaccine. Vaccine. 2025 Nov 14;66:127836. doi: 10.1016/j.vaccine.2025.127836. Epub 2025 Oct 14. PMID 41092804
- [Derived] Nogueira ML, Cintra MAT, Moreira JA, Patino EG, Braga PE, Tenorio JCV, de Oliveira Alves LB, Infante V, Silveira DHR, de Lacerda MVG, Pereira DB, da Fonseca AJ, Gurgel RQ, Coelho IC, Fontes CJF, Marques ETA, Romero GAS, Teixeira MM, Siqueira AM, Boaventura VS, Ramos F, Junior EE, de Moraes JC, Whitehead SS, Esteves-Jaramillo A, Shekar T, Lee JJ, Macey J, Kelner SG, Coller BG, Boulos FC, Kallas EG; Phase 3 Butantan-DV Working Group. Efficacy and safety of Butantan-DV in participants aged 2-59 years through an extended follow-up: results from a double-blind, randomised, placebo-controlled, phase 3, multicentre trial in Brazil. Lancet Infect Dis. 2024 Nov;24(11):1234-1244. doi: 10.1016/S1473-3099(24)00376-1. Epub 2024 Aug 5. PMID 39116904
- [Derived] Kallas EG, Cintra MAT, Moreira JA, Patino EG, Braga PE, Tenorio JCV, Infante V, Palacios R, de Lacerda MVG, Batista Pereira D, da Fonseca AJ, Gurgel RQ, Coelho IC, Fontes CJF, Marques ETA, Romero GAS, Teixeira MM, Siqueira AM, Barral AMP, Boaventura VS, Ramos F, Elias Junior E, Cassio de Moraes J, Covas DT, Kalil J, Precioso AR, Whitehead SS, Esteves-Jaramillo A, Shekar T, Lee JJ, Macey J, Kelner SG, Coller BG, Boulos FC, Nogueira ML. Live, Attenuated, Tetravalent Butantan-Dengue Vaccine in Children and Adults. N Engl J Med. 2024 Feb 1;390(5):397-408. doi: 10.1056/NEJMoa2301790. PMID 38294972